CLINICAL TRIAL: NCT04520490
Title: Brain Systems and Behaviors Underlying Response to Obesity Treatment in Children
Brief Title: Brain Activation and Satiety in Children 2
Acronym: BASIC2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Christian L Roth, MD, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00001984
Record Dates: First submitted 2020-07-31; First posted 2020-08-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exenatide once weekly extended-release (Active Comparator): Weekly subcutaneous injections of glucagon-like peptide (GLP)-1 agonist exenatide once weekly extended-release (2mg) for 24 weeks in randomized intervention.
  Interventions: Behavioral: Family Based Behavioral Treatment; Drug: Exenatide 2 mg [Bydureon]
- Matching placebo (Placebo Comparator): Weekly subcutaneous injections of placebo for 24 weeks.
  Interventions: Behavioral: Family Based Behavioral Treatment; Drug: Placebo

INTERVENTIONS:
Behavioral: Family Based Behavioral Treatment — Children with obesity accompanied by at least one parent or caregiver will attend 24 weekly sessions. Most sessions will be held via video-conference and include 25-30 min. meetings between an interventionist and each child/parent pair to individualize treatment, followed by separate child and parent group meetings lasting 40 - 45 min. A select few sessions will be held in-person between an interventionist and each child/parent pair with no group session. Parents will serve as primary agents of change for their child and for themselves. Training will focus on food and physical activity education, parenting around food and physical activity, and use of behavioral skills (e.g., self-monitoring, environmental control, contingency management). Intervention groups of 8-12 children/families will be initiated every 3-6 mos. in study yrs. 2-3.
Drug: Exenatide 2 mg [Bydureon] — Weekly injections of active drug.
  Other Names: Bydureon®
  Arms: Exenatide once weekly extended-release
Drug: Placebo — Weekly placebo injections
  Arms: Matching placebo

SUMMARY:
Childhood obesity and related long-term effects are serious public health problems, but not all children with obesity do well in treatment. This study will test a new combination of family-based behavioral treatment (FBT) with a drug intervention using a glucagon-like peptide-1 receptor agonist (GLP-1RA) exenatide once weekly extended-release (ExQW, Bydureon®) in order to improve obesity intervention outcomes in 10-12-year-old children.

DETAILED DESCRIPTION:
Using functional and structural magnetic resonance neuroimaging, this study will evaluate brain factors which could undermine treatment responses and long-term obesity intervention outcomes. Specific Aim 1 will test the effect of adding ExQW to FBT on change in BMI z-score over a total GLP-1RA treatment duration of 24 weeks and a subsequent 1-year observational follow-up period after treatment cessation. To provide mechanistic insight, Specific Aim 2 will test whether adding GLP-1RA intervention to FBT impacts neural activation by food cues. Finally, the proposed research will investigate the role of a cellular inflammatory process in the mediobasal hypothalamus-called gliosis-which might contribute to impaired hypothalamic function, attenuated satiety responsiveness, and potentially to worse weight management outcomes. Specific Aim 3 will test if hypothalamic gliosis is modified by FBT and/or FBT plus GLP-1RA in children and if its extent is related to immediate and/or long-term intervention outcomes.

Study Design: This double-blinded, randomized, placebo-controlled research study uses fMRI to characterize neural responses to a test meal before and at the end of FBT intervention, with vs. without additional GLP-1RA intervention. In addition, it uses structural MRI (sMRI) to test if MBH gliosis is reversible and/or associated with intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 10-12 years of age
* Male or female
* Ability and willingness to participate in study visits including fMRI scans, blood draws, and weekly injections;
* Parent willing to provide informed written consent and child willing to provide written assent;
* Child has BMI z-score >95th percentile. for age and sex;
* One parent that is obese or overweight (BMI >27 kg/m2); willingness of 1 parent (does not have to be the parent with obesity) to engage in weekly family-based weight control treatment delivered in English.

Exclusion Criteria:

* History of acute or chronic serious medical conditions;
* known diabetes mellitus or recent (6 mo.) history of anemia;
* Presence of any implanted metal or metal devices, including ferro-metallic surgical clips or orthodontic braces;
* Claustrophobia;
* Documented cognitive disorder, disruptive behavior, inability to participate in group sessions;
* Current use of medications known to alter appetite, body weight, or brain response
* Food intolerance to test meal (macaroni and cheese) or vegetarianism/veganism or severe food allergies.
* Known renal impairment (GFR<60 ml/min/1.73m2)
* History of gastroparesis, pancreatitis or gallstones (unless status post cholecystectomy);
* Family history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma;
* Known elevated calcitonin level at phone screening or increased measured calcitonin level at study visits;
* Untreated thyroid disorder or adrenal insufficiency;
* Use of weight loss medications (child participant) within 3 months of screening visit.
* Participating parent is pregnant

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Change of BMI z-score | Change from drug treatment randomization at week 8 of family-based behavioral treatment (FBT) to end of combined intervention (FBT + drug) at week 24 of FBT
  Body mass index (BMI) z-scores will be derived using CDC growth charts, using the LMS method, to allow for comparison of adiposity over time and across children who differ in age and sex.

SECONDARY OUTCOMES:
BMI z-score | Up to 12-months after ending treatment
  Change of body mass index (BMI) z-scores derived using CDC growth charts, using the LMS method, to allow for comparison of adiposity over time and across children who differ in age and sex.
Body composition | Change from Baseline to post-Family Based Behavioral Treatment at week 24 and post drug-treatment at week 32
  Changes in body composition as assessed using a bioelectrical impedance (BIA)
Indices of metabolic syndrome | Change from Baseline to post-Family Based Behavioral Treatment at week 24
  Changes of insulin resistance assessed by fasting insulin used for homeostasis model assessment of insulin resistance (HOMA-IR) using the formula insulin [mU/l] x glucose [mmol/l]) / 22.5
Meal induced chances in brain activation to visual food cues | Change from Baseline to post-Family Based Behavioral Treatment at week 24
  Change of brain response to visual food cues measured by functional magnetic resonance imaging in a priori regions of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No